CLINICAL TRIAL: NCT00662688
Title: Chemotherapy With or Without Preventive Anticoagulation for Metastatic Cancer of the Pancreas
Brief Title: Chemotherapy With or Without Dalteparin in Treating Patients With Metastatic Pancreatic Cancer
Acronym: PAM07
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitment prematurely stopped due to a lack of eligible patients.
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000593019; GERCOR-PAM07-D07-2; EUDRACT 2007-002115-59; EU-20837; PFIZER-GERCOR-PAM07-D07-2
Record Dates: First submitted 2008-04-18; First posted 2008-04-21 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Chemotherapeutic Agent Toxicity; Pancreatic Cancer; Thromboembolism
Keywords: thromboembolism; chemotherapeutic agent toxicity; adenocarcinoma of the pancreas; stage IV pancreatic cancer; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chemotherapy (Active Comparator): chemotherapy at investigator's discretion
  Interventions: Drug: Chemotherapy at the investigator's discretion
- dalteparin (Experimental): dalteparin: 5000 UI sub-cutaneous injection, from Day 1 to Day 28.
  Interventions: Drug: daltéparine; Drug: Chemotherapy at the investigator's discretion

INTERVENTIONS:
Drug: daltéparine
  Arms: dalteparin
Drug: Chemotherapy at the investigator's discretion

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Anticoagulants, such as dalteparin, may help prevent blood clots from forming in patients being treated with chemotherapy. It is not yet known whether gemcitabine is more effective when given alone or together with dalteparin and/or capecitabine in treating patients with pancreatic cancer.

PURPOSE: This randomized phase III trial is studying whether dalteparin prevents blood clots in patients with pancreatic cancer receiving treatment with different combinations of gemcitabine and capecitabine.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To demonstrate that preventive anticoagulation with dalteparin reduces the number of thromboembolic events.
* To determine the number of thromboembolic events occurring with preventive anticoagulation.

Secondary

* To determine survival without thrombotic event.
* To determine progression-free and overall survival.
* To determine time to response of tumor.
* To assess tolerance of these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center and WHO performance status (0-1 vs 2). Patients are randomized to 1 of 4 treatment arms.

* Arm A: Patients receive chemotherapy at investigator's discretion
* Arm B Patients receive chemotherapy at investigator's discretion and dalteparin In all arms, treatment repeats in the absence of disease progression or unacceptable toxicity.

Blood and plasma samples are obtained at baseline and periodically during study. Blood is examined for biomarkers, resistance to activated protein C, and mutations (Leiden V factor, mutation G20210A, and the factor II gene). Thrombin generation and factors VIIa and VIII are assessed in plasma.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas

  * Metastatic disease
  * Not amenable to treatment
  * No localized or locally advanced disease
* Measurable disease (metastatic or primary tumor) defined as ≥ 2 cm by CT scan or ≥ 1 cm by spiral CT scan or MRI
* No progressive thrombo-embolic disease
* No adenocarcinoma of the biliary tract or ampulla of Vater
* No known CNS metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy > 12 weeks
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Alkaline phosphatase < 5 times normal
* Bilirubin < 1.5 times normal
* Creatinine < 1.5 times normal
* Creatinine clearance < 30 mL/min
* Pain controlled or stabilized via analgesic therapy
* Affiliation with social security system
* Not pregnant or nursing
* No controlled or uncontrolled jaundice
* No contraindication to study drugs
* No cardiovascular accident (myocardial infarction, cerebral vascular accident) within the past 6 months
* No serious cardiac and/or respiratory disease
* No other cancer in the past 5 years except the following cancers, provided they have been completely resected:

  * Skin cancer
  * Localized melanoma
  * Carcinoma in situ of the cervix
* No history of thrombophilia
* No history of heparin-induced thrombocytopenia
* No uncontrolled or persistent hypercalcemia
* No psychological, familial, social, and/or geographical condition that precludes participation in the study

PRIOR CONCURRENT THERAPY:

* No prior hematologic therapy for metastatic disease
* No prior abdominal radiotherapy
* No concurrent corticosteroids as anti-emetic therapy
* No other concurrent anticoagulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Thromboembolic events | during study treatment
  number of thromboembolic events during anticoagulation treatment

SECONDARY OUTCOMES:
Progression-free survival | at 6 months
Overall survival | at one year
Tolerance of regimens | each cycle

CONTACTS AND LOCATIONS:
Overall Officials: Benoist Chibauldel, MD, Principal Investigator — Hopital Saint Antoine
Locations (6):
- France (6):
  - Centre Hospitalier de Meaux, Meaux
  - Centre Hospitalier Intercommunal Le Raincy - Montfermeil, Montfermeil
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Saint Antoine, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Foch, Suresnes

REFERENCES:
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539